CLINICAL TRIAL: NCT03873844
Title: Improving Thinking in Everyday Life: Pilot Study A
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Gitendra Uswatte, Professor, Department of Psychology, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-300002814
Record Dates: First submitted 2019-03-11; First posted 2019-03-14 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Impairment
Keywords: cognitive processing, transfer package
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Pilot study. Two baseline assessments precede intervention, which is followed by post-treatment testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CI Cognitive Therapy (Experimental): The treatment will have 2 components. The first component, Speed of Processing Training, is a computer game. Participants identify targets on the screen as rapidly as possible. The second component is a set of psychological techniques that will help participants apply the improvements from the game to carrying out tasks that rely on thinking in their daily life.
  Interventions: Behavioral: Speed of Processing Training; Behavioral: Transfer Package from CI Therapy

INTERVENTIONS:
Behavioral: Speed of Processing Training — Speed of Processing Training (SOPT). Speed of processing training involves trainer-guided practice of computer-based video "games." The "games" require the "player" to identify targets that are presented very briefly. SOPT has the primary aim of improving the fluid ability of mental processing speed such that trainees can process increasingly more information and increasingly more complex information over briefer periods of time. The training primarily involves practice with feedback. Trainers also offer suggestions, encouragement, and personalized modifications of difficulty for the trainee according to a specified protocol. At a display speed and task difficulty level tailored to their ability, trainees practice blocks of 16 trials. Trainees receive immediate feedback after each trial and see their total correct trials at the end of each block of trials. Trainers tell the trainees that their goal is to achieve performance of 10 to 12 correct trials for each training block.
Behavioral: Transfer Package from CI Therapy — Behavioral Contract. At the outset of treatment, the therapist negotiates a contract with the participant and caregiver, if one is available.Daily home diary. During treatment, the participants catalog the ADL and IADL for the part of the day spent outside the laboratory. Daily administration of the Cognitive Task Activity Log (CTAL). The CTAL collects information about attempts by the participant to complete ADL and IADL. Problem Solving. The therapist helps participants to think through any barriers to completing ADL and IADL independently. Home skill assignments during treatment. Participants are assigned on a written check-off sheet 10 specific ADL tasks. Home skill assignments after treatment. Toward the end of treatment, a written individualized post-treatment program is developed containing a list of up to 10 IADL for each day of the week. Post-treatment telephone contacts. Participants are contacted during the 12 month period after treatment to evaluate treatment outcomes.

SUMMARY:
This is a pilot study at the University of Alabama at Birmingham. The purpose of this initial study is to test how effective a new therapy is for improving participants ability to think, particularly how rapidly they process information that they receive from their senses, e.g., sight, hearing,… . The study will also test whether the new therapy improves how often and how well they are able to carry out tasks that rely on thinking in their daily life. The therapy will combine a computer game that ask participants to identify targets on the screen as rapidly as possible with a set of psychological techniques that will help to apply the improvements that are made in how rapidly participants process information as a result of the game to carrying out tasks that rely on thinking in your daily life.

DETAILED DESCRIPTION:
The purpose of this pilot study is to develop and test an intervention for slow processing of sensory input that not only increases the speed of processing but also produces improvement in how much and how well adults with this type of cognitive impairment carry out everyday tasks that rely on cognitive function. The intervention will combine Speed of Processing Training (SOPT) with a modified form of the Transfer Package from Constraint-Induced Movement therapy (CI therapy). SOPT has been shown to increase speed of processing in a variety of patient populations. The Transfer Package has been shown to produce transfer of gains from the treatment setting to everyday life when combined with training of arm use in the treatment in adults after stroke. The length of each treatment session will vary from 2 to 3.5 hours per day, the number of treatment days per week will range from 2 to 5, and the number of weeks of treatment will range from 2 to 10. Accordingly, the interval between testing occasions may change depending on the findings from initial pilot work. Total hours of treatment will not exceed 35. Ranges are given rather than precise values because part of the purpose of this pilot work is to decide, on a preliminary basis, what is the best schedule of delivery. In addition, four follow-up telephone calls will be conducted each week for the first month after the end of treatment. Then, a follow-up telephone call will be placed once a month for up to 11 months. These telephone calls will permit elements of the Transfer Package to be delivered remotely, helping the patient to transition from taking part in treatment to living their daily lives. Each telephone call will last 30 to 60 minutes. The outcomes that will be assessed are: speed of processing, performance of instrumental activities of daily living (IADL) that place demands on cognitive activity in the laboratory setting, and performance of IADL that place demands on cognitive activity outside the laboratory setting. There will be two baseline testing sessions, followed by post-treatment testing, and testing six months and 12 months after treatment. The two baseline testing sessions will be separated by a week, and will permit any changes observed after treatment to be compared to what takes place when no treatment is provided. In other words, the baseline testing sessions will provide a source of within-subject control. If a caregiver is available, the caregiver will be asked to complete CTAL interviews about the participant (see below) and will be invited to support the participant in following the Transfer Package elements of the treatment (see below). Repeated measures analysis of variance models will be used to evaluate if statistically significant improvements take place as a result of treatment.

ELIGIBILITY:
Inclusion Criteria:

* impairment in speed of processing. This will determined by a time greater than 100 ms on Task 2 and greater than 300 ms on Task 3 of the Useful Field of View test
* substantial impairment in performance of daily activities. This will be determined by a score of at most 2.5 on the Cognitive Task Activity Log
* presence of a stroke, including vascular dementia, TBI, or cognitive impairment due to other causes
* at least 3 months since brain injury for participants with stroke or TBI
* 18 years or older
* medically stable
* sufficiently fit, from both a physical and mental health perspective, to take part in study
* adequate sight and hearing to complete UFOV test
* adequate thinking skills, i.e., ability to follow directions, retain information, to complete UFOV and CTAL, per judgement of the screener
* reside in the community (as opposed to a hospital or skilled nursing facility)
* able to travel to laboratory on multiple occasions

Exclusion Criteria:

- n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Cognitive Task Activity Log (CTAL) | Change from Day 0 to Day 28
  The CTAL collects information about attempts by the participant to complete activities of daily living (ADL) and instrumental ADL (IADL).

SECONDARY OUTCOMES:
Useful Field of View (UFOV) | Change from Day 0 to Day 28
  This test is very similar to the SOPT training program (see paragraph on SOPT in Treatment section above). The UFOV Assessment quantifies how rapidly test takers process sensory input. It is well validated test, that is used widely. It has been adopted by Federal and State agencies and insurance companies to assess fitness to drive, which is closely related to speed of processing.

OTHER OUTCOMES:
Timed Instrumental Activities of Daily Living | Change from Day 0 to Day 28
  This test measures how rapidly participants can complete five timed tasks that simulate everyday instrumental activities of daily living in the laboratory. Tasks are: 1. finding a telephone number of a specific individual in the telephone directory, 2. finding and correctly counting out 37 cents from a group of coins, 3. finding and reading the ingredients on a food can label, 4. finding two food items in an array of food items simulating a crowded pantry shelf, and 5. finding and reading the directions on a medicine container. The tester records the time required to complete each task. If the participant does not complete the task within the preset time limit, testing for that particular task discontinues. The tester adds a penalty to completion time for the tasks completed with minor errors, transforms the times for each of the tasks into z-scores, and calculates the average of the transformed scores. This test has been validated and was used in a multi-site clinical trial test

CONTACTS AND LOCATIONS:
Overall Officials: Edward Taub, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No
This is pilot study. A major purpose of this study is simply to develop the intervention. Sharing individual data is premature.